CLINICAL TRIAL: NCT03774472
Title: Phase I/II Safety and Efficacy Study of Autophagy Inhibition With Hydroxychloroquine to Augment the Antiproliferative and Biological Effects of Pre-Operative Palbociclib Plus Letrozole for Estrogen Receptor-Positive and HER2-Negative Breast Cancer
Brief Title: Hydroxychloroquine, Palbociclib, and Letrozole Before Surgery in Treating Patients With Estrogen Receptor Positive, HER2 Negative Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0071; NCI-2018-01050 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0071 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-12-07; First posted 2018-12-13 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: interventions — Hydroxychloroquine; Letrozole; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (hydroxychloroquine, palbociclib, letrozole) (Experimental): PHASE I: Patients with advanced, metastatic (stage IV) breast cancer receive hydroxychloroquine PO QD, palbociclib PO QD, and letrozole PO QD on days 1-28. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  PHASE II: Patients with early stage (stage I-III) breast cancer receive hydroxychloroquine PO QD on days 15-28 of cycle 1 and on days 1-28 of subsequent cycles. Patients also receive palbociclib PO QD, and letrozole PO QD on days 1-28, followed by standard of care surgery at week 5. If there is a proliferative benefit with CCCA by biopsy at 4 weeks, cycles may repeat every 28 days for up to 20-24 weeks in the absence of disease progression or unacceptable toxicity, followed by standard of care surgery during weeks 20-24.
  Interventions: Drug: Hydroxychloroquine; Drug: Letrozole; Drug: Palbociclib

INTERVENTIONS:
Drug: Hydroxychloroquine — Given PO
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara
Drug: Palbociclib — Given PO
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991

SUMMARY:
This phase I/II trial studies the side effects and best dose of hydroxychloroquine when given together with palbociclib and letrozole before surgery in treating patients with estrogen receptor positive, HER2 negative breast cancer. Hydroxychloroquine is a substance that decreases immune responses in the body. Palbociclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Estrogen can cause the growth of breast cancer cells. Drugs, such as letrozole, may lessen the amount of estrogen made by the body. Giving hydroxychloroquine, palbociclib, and letrozole before surgery may work better than palbociclib and letrozole in treating patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of adding hydroxychloroquine (HCQ) to continuous low dose palbociclib and letrozole and to determine the recommended phase II dose (RP2D) for hydroxychloroquine (HCQ) for the subsequent Phase II study. (Phase I) II. To determine the dose responsiveness of 2 dose levels (400 mg and recommended phase II dose [RP2D]) of hydroxychloroquine added to low dose palbociclib and letrozole on pre and post HCQ breast tumor proliferation index (Ki67), autophagy, senescence and cell cycle control. (Phase II, Part I) III. To determine whether hydroxychloroquine added to low dose palbociclib and letrozole can increase the proportion of patients whose tumors achieve complete cell cycle arrest (CCCA, defined as the Ki67 =< 2.7%) comparing T2 to T1. (Phase II, Part II)

SECONDARY OBJECTIVES:

I. To determine the response rate and clinical benefit rate at 8 weeks of the assigned dose of hydroxychloroquine (HCQ) plus continuous low dose palbociclib and letrozole. (Phase I) II. Determine longer term clinical tumor responsiveness (tumor volume) and tumor biomarker indices (for patients who have extended pre-operative therapy, maximum 24 weeks). (Phase II, Part I) III. Perform exploratory studies on blood-based tumor protein, deoxyribonucleic acid (DNA) and ribonucleic acid (RNA) biomarkers with a focus on pathways of cell proliferation, autophagy, senescence and cell cycle control. (Phase II, Part I) IV. To determine the impact of adding hydroxychloroquine to low dose palbociclib and letrozole on breast tumor indices of proliferation, autophagy, senescence, cell cycle control and other intersecting pathways. (Phase II, Part II) V. Determine longer term clinical tumor responsiveness and tumor biomarkers indices (for patients who have extended pre-operative therapy, maximum 24 weeks). (Phase II, Part II) VI. To determine the dose responsiveness of HCQ (400 mg vs. RP2D) on the primary (proportion with CCCA) and secondary clinical/biological endpoints. (Phase II, Part II) VII. To perform exploratory studies on blood-based tumor protein, DNA and RNA biomarkers. (Phase II, Part II) VIII. Obtain additional safety information for the combination of low dose palbociclib, letrozole and hydroxychloroquine. (Phase II, Part II)

OUTLINE: This is a phase I, dose-escalation study of hydroxychloroquine followed by a phase II study.

PHASE I: Patients with advanced, metastatic (stage IV) breast cancer receive hydroxychloroquine orally (PO) once daily (QD), palbociclib PO QD, and letrozole PO QD on days 1-28. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients with early stage (stage I-III) breast cancer receive hydroxychloroquine PO QD on days 15-28 of cycle 1 and on days 1-28 of subsequent cycles. Patients also receive palbociclib PO QD, and letrozole PO QD on days 1-28, followed by standard of care surgery at week 5. If there is a proliferative benefit with complete cell cycle arrest (CCCA) by biopsy at 4 weeks, cycles may repeat every 28 days for up to 20-24 weeks in the absence of disease progression or unacceptable toxicity, followed by standard of care surgery during weeks 20-24.

After completion of study treatment, patients are followed up within 30 days or every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Diagnosis of estrogen positive breast cancer, estrogen receptor-positive and HER2-negative by American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Postmenopausal defined by: a. Age >= 55 years and 1 year or more of amenorrhea b. Age < 55 years and 1 year or more of amenorrhea with luteinizing hormone (LH) and/or follicle stimulating hormone (FSH) levels in the postmenopausal range c. Age < 55 with prior hysterectomy but intact ovaries with LH and/or FSH levels in the postmenopausal range d. Chemotherapy or medically induced ovarian suppression with 1 year or more of amenorrhea and with LH and/or FSH levels in the postmenopausal range e. Status after bilateral oophorectomy (>= 28 days prior to first study treatment)
* Absolute neutrophil count (ANC) >= 1500 cells/ul
* Platelet count >= 100,000/ul
* Serum creatinine concentration < 1.5 x upper limit of normal (ULN)
* Bilirubin level < 1.5 x ULN
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 x ULN
* Alkaline phosphatase =< 2.5 ULN
* Metastatic cohorts (Phase I): Diagnosis of stage IV estrogen positive breast cancer, estrogen receptor-positive and HER2-negative by ASCO/CAP criteria
* Metastatic cohorts (Phase I): Must be a candidate for treatment with CDK4/6 inhibitor and hormonal therapy with an aromatase inhibitor as standard of care
* Metastatic cohorts (Phase I): No prior exposure to CDK 4/6 inhibitors
* Neoadjuvant cohorts (Phase II): Diagnosis of stage I-III estrogen positive breast cancer, estrogen receptor-positive and HER2-negative by ASCO/CAP criteria. If stage I, clinical tumor size must be >= 1.5 cm
* Neoadjuvant cohorts (Phase II): Baseline tumor Ki67 > 5%
* Neoadjuvant cohorts (Phase II): Surgical candidate and appropriate for pre-operative endocrine therapy

Exclusion Criteria:

* Prior exposure to CDK 4/6 inhibitor therapy
* History of retinal disease or active visual disturbances (normal baseline study-specified retinal exam required)
* Acute illness, including infections requiring medical therapy, known bleeding diathesis or need for anticoagulation
* Treatment with any of the following medications within 4 weeks before the baseline diagnostic biopsy is taken: a. Oral estrogens, including hormone replacement therapy (but prior depot estrogen use not allowed). b. Investigational agents (or 5 half-lives, whichever is longer)
* Required concomitant use of any drug that is a strong CYP3A inhibitor or inducer
* Psychological, familial, sociological or geographical conditions that do not permit compliance with the study protocol
* Life expectancy of less than 6 months
* Pregnancy, lactation or planning to be pregnant.
* Neo-adjuvant cohorts (Phase II): Prior therapy for breast cancer (medical, surgical or radiation therapy)
* Neo-adjuvant cohorts (Phase II): Clinical T4 disease
* Neo-adjuvant cohorts (Phase II): Inoperable or metastatic breast cancer based on standard evaluation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debasish Tripathy, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Raghavendra AS, Kettner NM, Kwiatkowski D, Damodaran S, Wang Y, Ramirez D, Gombos DS, Hunt KK, Shen Y, Keyomarsi K, Tripathy D. Phase I trial of hydroxychloroquine to enhance palbociclib and letrozole efficacy in ER+/HER2- breast cancer. NPJ Breast Cancer. 2025 Jan 26;11(1):7. doi: 10.1038/s41523-025-00722-1. PMID 39865083
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- HCQ at 400mg; HCQ at 600mg; HCQ at 800mg: PHASE I: Patients with advanced, metastatic (stage IV) breast cancer receive hydroxychloroquine PO QD, palbociclib PO QD, and letrozole PO QD on days 1-28. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | HCQ at 400mg | HCQ at 600mg | HCQ at 800mg
Started | 4 | 5 | 6
Completed | 3 | 3 | 6
Not Completed | 1 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Progression prior to 4 weeks | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- HCQ at 400 mg; HCQ at 600 mg; HCQ at 800 mg: PHASE I: Patients with advanced, metastatic (stage IV) breast cancer receive hydroxychloroquine PO QD, palbociclib PO QD, and letrozole PO QD on days 1-28. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | HCQ at 400 mg | HCQ at 600 mg | HCQ at 800 mg | Total
Number analyzed (Participants) | 4 | 5 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 6 | 15
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 6 | 15
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 6 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 2 | 4 | 6 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (Phase I)
Description: Incidence of adverse events (Phase I) [Time Frame: Up to 30 days post-treatment] Assessed continuously using Common Terminology Criteria for Adverse Events version 4.03, with physical examination and laboratory assessments.
Time Frame: Up to 5 years and 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | HCQ at 400 mg | HCQ at 600 mg | HCQ at 800 mg
Number analyzed (Participants) | 3 | 3 | 6
Participants | 3 | 3 | 6

2. Secondary Outcome: Recommended Phase II Dose for HCQ
Description: Phase I portion in the metastatic setting is to determine the safety of adding HCQ to continuous low dose palbociclib and letrozole and to determine the recommended phase II dose for HCQ for the subsequent Phase II study.
Time Frame: Up to 5 years and 4 months
Measure: Number; unit: mg/day
Groups:
- Experimental: Treatment (Hydroxychloroquine, Palbociclib, Letrozole): PHASE I: Patients with advanced, metastatic (stage IV) breast cancer receive hydroxychloroquine PO QD, palbociclib PO QD, and letrozole PO QD on days 1-28. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
Arm/Group | Experimental: Treatment (Hydroxychloroquine, Palbociclib, Letrozole)
Number analyzed (Participants) | 12
mg/day | 800

3. Secondary Outcome: Clinical Benefit Rate at 8 Weeks
Description: The secondary objective is to determine the response rate and clinical benefit rate at 8 weeks of the assigned HCQ dose plus continuous low dose palbociclib and letrozole.
Time Frame: Up to 5 years and 4 months
Measure: Number; unit: percentage of participants
Arm/Group | HCQ at 400 mg | HCQ at 600 mg | HCQ at 800 mg
Number analyzed (Participants) | 3 | 3 | 6
percentage of participants | 100 | 66.6 | 100

ADVERSE EVENTS:
Time Frame: Up to 5 years and 4 months
Arm/Group | HCQ at 400mg | HCQ at 600mg | HCQ at 800mg
All-Cause Mortality (participants affected / at risk) | 2/4 | 0/4 | 2/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCQ at 400mg (N=4) | HCQ at 600mg (N=4) | HCQ at 800mg (N=6)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 3 (3)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 5 (5)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT03774472/Prot_SAP_000.pdf